CLINICAL TRIAL: NCT06497361
Title: Safety and Efficacy of PRG-2311 (CD19/BCMA-targeting CAR-T Cells) for Refractory Lupus Nephritis and IgG4-Related Disease
Brief Title: Safety and Efficacy of PRG-2311 for Refractory Lupus Nephritis and IgG4-Related Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lingli Dong, Professor of the department of rheumatology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Tongji Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S114
Record Dates: First submitted 2024-06-27; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Lupus Nephritis; IgG4-related Disease
MeSH Terms: conditions — Lupus Nephritis; Immunoglobulin G4-Related Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T cells therapy (Experimental): The study was divided into two phases: dose exploration phase and dose extension phase. Three dose levels (35×10^6 CAR-T, 100×10^6 CAR-T, 300×10^6 CAR-T) were planned for the dose-exploration phase, and 3 to 6 LN or IgG4-RD subjects were included in each dose group. When 1 out of 3 subjects in a dose group showed DLT, 3 subjects were re-enrolled at that dose level. If DLT occurs in ≥2 of 6 subjects, dose reduction or study termination should be considered.
  The safe and effective fixed dose of PRG-2311 was determined through the dose-exploration phase, and after evaluation by the investigators, the dose-expansion phase was conducted, in which an additional 3-6 subjects were included in the safe and effective fixed dose for each of the two indications (Lupus Nephritis and IgG4-Related Disease) to further determine the safety and efficacy of this dose for each indications.
  Interventions: Biological: PRG-2311

INTERVENTIONS:
Biological: PRG-2311 — PRG-2311 (CD19/BCMA-targeting CAR-T Cells)

SUMMARY:
A Clinical Study on the Safety and Effectiveness of CD19/BCMA Chimeric Antigen Receptor T Cells in the Treatment of Refractory Lupus Nephritis and IgG4-Related Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. If the kidneys are involved, estimate the glomerular filtration rate (eGFR) to be ≥ 15 mL/minute/1.73 m2;
3. The following test values within 3 days before the collection of mononuclear cells meet the following standards:

   1. Absolute lymphocyte count: ≥ 0.5 × 10 ^ 9/L [The use of granulocyte colony-stimulating factor (G CSF) is allowed, but subjects are not allowed to receive this supportive treatment within 7 days before the screening period laboratory examination];
   2. Absolute neutrophil count: ≥ 1.0 × 10 ^ 9/L [The use of granulocyte colony-stimulating factor (G-CSF) is allowed, but subjects are not allowed to receive this supportive treatment within 7 days before the screening period laboratory examination];
   3. Platelets: Subject platelet count ≥ 50 × 10 ^ 9/L (subjects are not allowed to receive blood transfusion support within 7 days before the screening period laboratory examination);
   4. Hemoglobin: ≥ 8.0 g/dL (allowing the use of recombinant human erythropoietin) [subjects have not received red blood cell (RBC) infusion within 7 days prior to the screening period laboratory examination];
   5. Creatinine clearance rate: (CrCl) or glomerular filtration rate (GFR) (Cockcroft Gault formula) ≥ 30 mL/min;
   6. Total bilirubin (serum): Total bilirubin (serum) ≤ 1.5 × ULN; Blood bilirubin>1.5 × Gilbert subjects from ULN can be enrolled with the consent of the sponsor AST and ALT: ≤ 3.0 × ULN;
   7. Plasma prothrombin time (PT), international standardized ratio (INR), partial prothrombin time (APTT): PT ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN, INR ≤ 1.5 × ULN Willing to sign an informed consent form.
4. Fertile men and women of childbearing age must agree to use effective contraception from the time they sign an informed consent and up to 1 year after the study drug is used. Blood pregnancy tests for women of reproductive age at the time of screening and before cell infusion must be negative.
5. The patients or their guardians agree to participate in the clinical study and sign the informed consent, indicating that they understand the purpose and procedure of the clinical study and are willing to participate in the study.

   * for refractory LN

     1. According to the 2019 American Society of Rheumatology (ACR) criteria, diagnosed with systemic lupus erythematosus, within 6 months prior to infusion, confirmed by renal tissue biopsy according to the 2003 International Society of Nephrology (ISN)/Society of Nephropathology (RPS) criteria as active, proliferative lupus nephritis (LN), type III or IV, or type III/IV combined with type V, or type V. And have received standard treatment that is ineffective or relapses after disease remission.
     2. Positive anti-nuclear antibodies (ANA) and/or anti-dsDNA antibodies during the screening period.
     3. The SLE Disease Activity Index (SLEDAI-2000) score during the screening period is ≥ 8. SLEDAI-2000 clinical score ≥ 6 points, but low complement and/or anti ds-DNA positivity can be selected.
   * for refractory IgG4-RD

     1. According to the 2019 ACR/EULAR criteria, diagnosed with IgG4-RD;
     2. The clinical manifestations were recurrent or refractory IgG4-RD;
     3. IgG4-RD response index (RI) ≥2, the disease is in the active stage;
     4. meet the clinical phenotype of Mikulitz/systemic

Exclusion Criteria:

Subjects who meet any of the following criteria should be excluded from this study:

1. Pregnant or lactating women;
2. A history of malignant tumors within 5 years （①Carcinoma in situ of the cervix that has undergone curative treatment for more than 12 months prior to screening, ②Basal cell or squamous cell carcinoma of the skin that has been treated therapeutically, ③ Prostate cancer that has been treated with radical prostatectomy or curative radiation therapy for more than 3 years prior to screening has no known recurrence and is not currently receiving treatment；④have had surgery for thyroid cancer, and have not evidence of active disease）;
3. Received any B-cell depletion biologic therapy (for example, rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab, etc) in the 6 months prior to CAR-T reinfusion, unless B-cell recovery was demonstrated;
4. Received immunosuppressant therapy within 3 days prior to CAR-T reinfusion, or systemic corticosteroid therapy (>10 mg/ day of prednisone or equivalent doses of other corticosteroids) within 3 days prior to CAR-T reinfusion;
5. Received live vaccine or live therapeutic STDS within 2 weeks prior to screening;
6. The presence of chronic and active hepatitis B (except for HBV DNA testing below 500IU/ml), hepatitis C (HCV), human immunodeficiency virus (HIV) infection, or syphilis infection;
7. With an active infection that requires intravenous antibiotics or hospitalization;
8. Obvious evidence of cardiovascular disease as follows: a N-terminal B-type natriuretic peptide (NT proBNP)>8500ng/L; b. The New York Heart Association (NYHA) classifies heart failure as Grade IV; c. Patients who received hospitalization for unstable angina or myocardial infarction within 6 months prior to the first administration, or patients who received percutaneous cardiac intervention and received the most recent stent placement within 6 months or coronary artery bypass grafting within 6 months;
9. People who have a known allergy, hypersensitivity, intolerance, or contraindication to any component of PRG-2311 or the drugs that may be used in the study, including fludarabine, cyclophosphamide, tolumab, or albumin, or who have had a prior severe allergic reaction;
10. Patients with other conditions determined by the investigator to be unsuitable for lymphocyte clearance or cell infusion, or who are otherwise unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Safe dose of PRG-2311 infusion | Up to 24 months after PRG-2311 infusion
  To evaluate the safe dose of PRG-2311 infusion, 3 dosage group were designed in this trial, they are 35×10^6 CAR-T, 100×10^6 CAR-T, and 300×10^6 CAR-T
Occurrence of AE after PRG-2311 infusion | Up to 24 months after PRG-2311 infusion
  To evaluate the occurrence of AE after PRG-2311 infusion based on CTCAE v5.0

SECONDARY OUTCOMES:
LN: Changes of SLE disease activity Index (SLEDAI-2000) score | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  SLEDAI-2000 is the most commonly used SLE assessment scale. A total of 24 items, the total score is 105 points, scores ≤6 points indicates mild activity, ≥7 but ≤12 is classified as moderate activity, >12 is classified as severe activity.
LN: Changes of FACIT score | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  FACIT score is used to assess the fatigue status of patient
LN: Changes of PGA score | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  PGA score is used to assess the disease activity status of patient by physician
LN: Changes of UPCR | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  UCPR: urinary protein creatinine ratio (ug/mg)
LN: Changes of eGFR | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  eGFR : estimated glomerular filtration rate (ml/min/1.73m^2)
LN: overall response rate (complete or partial renal response | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  complete renal response rate or partial renal response rate
IgG4-RD: time to disease relapse | Up to 24 months after PRG-2311 infusion
  Definition:The number of days between the date of CAR-T infusion and the date of IgG4-RD recurrence determined by a clinical professional physician during the follow-up period
IgG4-RD: changes in the proportion of patients with improved disease activity (IgG4-RD RI) | Baseline,1st month, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  IgG4-RD (IgG4-RD RI) responder index is the most commonly used IgG4-RD assessment scale
IgG4-RD: The annual relapse rate | Up to 24 months after PRG-2311 infusion
  The annual recurrence rate
IgG4-RD: The proportion of patients achieved a complete response at week 52 | 24 months after cell infusion
  The proportion of complete response
PK: the feature of copy numbers of CAR-Cmax | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Cmax
PK: the feature of copy numbers of CAR-Tmax | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Tmax
PK: the feature of copy numbers of CAR-AUC0-28d | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Cmax、Tmax、AUC0-28d、AUC0-90d、T last of the copy numbers of CAR
PK: the feature of copy numbers of CAR-AUC0-90d | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  AUC0-90d
PK: the feature of copy numbers of CAR-T last of the copy numbers of CAR | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  T last of the copy numbers of CAR
PK: changes of the proportion of CAR-T cells to T cells | Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28, 2nd month, 3rd month
  Flow cytometry is used to detect the proportion of CAR-T cells to T cells.
PD: changes of the levels of plasma sBCMA, IgG, IgA, IgM, complement C3 and C4 | Screening period, Baseline, Day 14, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Immunology-related index
PD: changes of pathogenic antibody titers | Screening period, Baseline, Day 14, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Changes of ANA, anti-JO1, anti-SSA, anti-SSB, anti-Ro52, anti-centromerin B, anti-histone, anti-rRNP, anti-Scl70, anti smith, anti-ul-RNP and anti-dsDNA antibody titers in peripheral blood (only for enrolled lupus nephritis patients), and changes of IgG1, IgG2, IgG3, IgG4, and IgE (only for enrolled IgG4-RD patients)
PD: changes of immunoinflammation related laboratory indices | Screening period, Baseline, Day 2, Day 6, Day 10, Day 14, Day 21, Day 28 after cell infusion
  Changes of laboratory indices related to immune responses and inflammation in peripheral blood, including ESR, hsCRP, LDH, and serum cytokines
PD: changes of T and B lymphocyte subpopulations in peripheral blood | Screening period, Baseline, Day 14, Day 28, 2nd month, 3rd month, 6th month, 9th month, 12th month, 18th month, and 24th month after cell infusion
  Changes of lymphocyte subgroup in peripheral blood
BCMA expression levels of memory B cells and plasma blast cells | Screening period, baseline, Day 14, Day 28, month 2, month 3, month 6, month 9, month 12 and month 24
  BCMA expression levels of memory B cells and plasma blast cells in peripheral blood
Single cell sequencing | Screening period, 3 months after cell infusion (or B cell recovery stage), or depending on the investigator's assessment
  Single cell sequencing of peripheral blood T cells, B cells and CAR-T
The change of national planning vaccine antibody levels | Screening period, 3 months after cell infusion
  To evaluate the effect of CAR-T clearance of B cell on immunological protection after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Lingli Dong, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No